CLINICAL TRIAL: NCT05950191
Title: LLIN Evaluation in Uganda Project (LLINEUP3): Impact of Long-lasting Insecticidal Nets (LLINs) Treated With Chlorfenapyr Plus Pyrethroid vs LLINs Treated With Piperonyl Butoxide Plus Pyrethroid on Malaria Incidence in Uganda: a Cluster-randomised Trial
Brief Title: LLIN Evaluation in Uganda Project (LLINEUP3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Infectious Diseases Research Collaboration, Uganda (Other); Ministry of Health, Uganda (Other Government); Against Malaria Foundation (Unknown); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LLINEUP3; U19AI089674 (NIH)
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Malaria
Keywords: long lasting insecticidal nets with chlorfenapyr-pyrethroid; long lasting insecticidal nets with with PBO-pyrethroid
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Cluster-randomised trial to evaluate the impact of LLINs distributed in Uganda through the 2023 national universal coverage campaign. A cluster has been defined as the target area surrounding an MRC. A total of 24 clusters will be included in the study, covering 20 moderate-high malaria burden districts in Uganda. Clusters have been randomised in a 1:1 ratio to receive one of two types of LLINs: (1) chlorfenapyr-pyrethroid LLINs (PermaNet Dual, n=12) or (2) PBO-pyrethroid LLINs (PermaNet 3.0, n=12).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PermaNet Dual (Experimental): long lasting insecticidal nets with chlorfenapyr-pyrethroid
  Interventions: Other: long lasting insecticidal nets with chlorfenapyr-pyrethroid (PermaNet Dual); Behavioral: Social Behavior Change Communication
- PermaNet 3.0 (Active Comparator): long lasting insecticidal nets with PBO-pyrethroid
  Interventions: Other: long lasting insecticidal nets with PBO-pyrethroid (PermaNet); Behavioral: Social Behavior Change Communication

INTERVENTIONS:
Other: long lasting insecticidal nets with chlorfenapyr-pyrethroid (PermaNet Dual) — Next-generation bed net combining insecticides with different modes of action
  Arms: PermaNet Dual
Other: long lasting insecticidal nets with PBO-pyrethroid (PermaNet) — Next-generation bed net combining an insecticide with a synergist
  Arms: PermaNet 3.0
Behavioral: Social Behavior Change Communication — The NMCD and other stakeholders will take the lead on Social Behaviour Change Communication (SBCC). SBCC activities will use digital and other platforms, including the following: (1) LLIN launch at the World Malaria Day celebrations; (2) regional in-person advocacy meetings; (3) mass media platforms (for advertisements, mini skits, DJ mentions, radio spots, interactive talks); (4) social media platforms; (5) VHTs; (6) operation hotlines and toll-free call centres; (7) community mobilisation (megaphones); and (8) use of appropriate information, education, and communication materials. Communication will include messages about malaria, and use, care, repair and repurposing of bed nets.

SUMMARY:
In Uganda, the National Malaria Control Division (NMCD) and implementing partners are planning to deliver long-lasting insecticidal nets (LLINs) nationwide, through a mass distribution campaign in 2023. LLINs will be distributed free-of-charge to all Ugandan households, aiming to achieve universal coverage. LLINs treated with a pyrethroid insecticide plus chlorfenapyr (PermaNet Dual, Vestergaard) and LLINs treated with a pyrethroid insecticide plus PBO (PermaNet 3.0, Vestergaard) will be distributed as part of this distribution campaign, presenting an opportunity to rigorously evaluate and compare these two LLINs at scale across Uganda. In collaboration with the MOH, this cluster-randomised trial will compare the impact of LLINs combining chlorfenapyr with a pyrethroid to LLINs combining PBO with a pyrethroid into Uganda's 2023 LLIN distribution campaign, as was done successfully at the time of the last LLIN distribution campaign conducted in 2020-21. A major strength of this trial is the use of malaria incidence as the primary outcome measure. Incidence of malaria, defined as the number of symptomatic cases of malaria occurring in a population at risk over time, is the gold standard for assessing malaria burden. However, cluster-randomised trials using malaria incidence as the primary outcome typically involve study cohorts and are very expensive and logistically challenging. The novel approach for measuring malaria incidence is to utilize data collected routinely at health facilities. By defining target areas around health facilities and collecting data on the location of residence of patients diagnosed with malaria, this study will be able to generate longitudinal measures of malaria incidence at an unprecedented scale across Uganda as done in the LLINEUP2 trial (NCT04566510). These results will inform policies and programmes for malaria and potentially provide evidence to support widescale deployment of dual AI chlorfenapyr-pyrethroid LLINs. This study, the first evaluating PermaNet Dual LLINs, will also provide evidence for a second in class chlorfenapyr net, a potential tool to be added to the malaria control tool kit.

DETAILED DESCRIPTION:
This is a cluster-randomised trial to evaluate the impact of long-lasting insecticidal nets (LLINs) distributed in Uganda through the 2023 national universal coverage campaign. A cluster has been defined as the target area surrounding an MRC. A total of 24 clusters will be included in the study, covering 20 moderate-high malaria burden districts in Uganda. Clusters have been randomised in a 1:1 ratio to receive one of two types of LLINs: (1) chlorfenapyr-pyrethroid LLINs (PermaNet Dual, n=12) or (2) PBO-pyrethroid LLINs (PermaNet 3.0, n=12). The intervention, including delivery of the LLINs and social and behaviour change communication (SBCC), will be led by the Ugandan NMCD and other stakeholders. Currently, LLINs are scheduled to be distributed in the study areas during waves 5 and 6 from September to October 2023 as part of the national LLIN distribution campaign. The evaluation of the intervention will include: 1) health facility surveillance at the participating MRCs to generate continuous estimates of malaria incidence for each MRC target area; 2) cross-sectional community surveys at 12- and 24-months post-LLIN distribution to gather information on parasite prevalence, anaemia prevalence, net ownership, coverage, and use, 3) entomology surveys at 12 and 24 months to gather information on vector density. The primary outcome of the trial will be malaria incidence as estimated using the health facility surveillance.

ELIGIBILITY:
Household Survey

Inclusion Criteria:

1. At least one adult aged 18 years or older present
2. Adult is a usual resident who slept in the sampled household on the night before the survey
3. Agreement of the adult resident to provide informed consent for the household and entomology survey

Exclusion Criteria:

1. Dwelling destroyed or not found
2. Household vacant
3. No adult resident home on more than 3 occasions

Clinical Survey

Inclusion Criteria:

1. Usual resident who was present in the sampled household on the night before the survey
2. Agreement of adult or parent/guardian (of children) to provide informed consent
3. Agreement of child aged 8 years or older to provide assent

Exclusion Criteria:

1. Resident not home on day of survey

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 215903 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Number of cases of laboratory-confirmed malaria diagnosed at the MRC among patients residing in the target area | 24-months follow up
  malaria incidence: number of cases divided by the total population of the target area

SECONDARY OUTCOMES:
Prevalence of parasitaemia | 24-months following LLIN distribution
  Proportion of blood smears positive for parasites by microscopy in individuals of all ages at the time of cross-sectional surveys
Prevalence of anemia | 24-months following LLIN distribution
  Proportion of children aged 2-4 years with haemoglobin < 11 g/dL at the time of cross-sectional surveys
Proportion of households that owned at least one LLIN | 24-months following LLIN distribution
  Proportion of households with at least one LLIN at the time of cross-sectional surveys
Proportion of households that owned at least one LLIN for every two occupants | 24-months following LLIN distribution
  Proportion of households with at least one LLIN per every two occupants at the time of cross-sectional surveys
Proportion of household residents who slept under an LLIN the previous night | 24-months following LLIN distribution
  Proportion of households residents who report sleeping under LLIN the previous night at the time of cross-sectional surveys
Number of female anopheles mosquitoes collected per household at the time of cross-sectional surveys | 24-months following LLIN distribution
  Vector density

CONTACTS AND LOCATIONS:
Overall Officials: Moses Kamya, MBChB, MMed, PhD, Principal Investigator — Makerere University; Infectious Diseases Research Collaboration; Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No